CLINICAL TRIAL: NCT04887935
Title: Pilot Clinical Trial of Neoadjuvant SGLT2 Inhibition in Localized Prostate Cancer
Brief Title: Neoadjuvant SGLT2 Inhibition in Localized Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202107070
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Cancer of Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Dapagliflozin (Experimental): * Dapagliflozin will be initiated once daily approximately 6 weeks prior to planned prostatectomy
  * Dapagliflozin will be given at 10 mg by mouth once daily for 4 weeks (days 1-28) prior to prostatectomy.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — -The 10 mg dose is reflective of current clinical practice for diabetes and heart failure
  Other Names: Farxiga

SUMMARY:
This is a pilot study of the tolerability and safety of neoadjuvant dapagliflozin for patients with unfavorable intermediate, high-risk, or very high-risk prostatic adenocarcinoma prior to radical prostatectomy. The primary hypothesis is that four weeks of daily dapagliflozin prior to surgery is well-tolerated and safe to use in this patient population. The investigators also hypothesize that dapagliflozin will be efficacious in resulting in tumor shrinkage on pre-operative imaging and will result in tumor necrosis at prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed localized prostatic adenocarcinoma. Patients with primarily neuroendocrine/small cell histology will be excluded.
* Patients with prostatic adenocarcinoma in one of the following risk groups as defined by NCCN criteria:

  * Unfavorable intermediate risk. Intermediate risk is defined as having no high-risk or very high-risk factors and having at least one of the following intermediate risk factors (IRFs):

    * cT2b-cT2c
    * Grade Group 2 or 3
    * PSA 10-20 ng/mL
    * Unfavorable intermediate risk additionally must have one or more of the following:

      * 2 or 3 IRFs
      * Grade Group 3
      * ≥50% biopsy cores positive (eg, ≥ 6 of 12 cores) OR
  * High-risk, which is defined as not meeting very high-risk criteria and having at least one of the following high-risk features:

    * cT3-cT4
    * Grade Group 4 or 5
    * PSA > 20 ng/mL OR
  * Very high-risk, which is defined as meeting at least two of the following criteria:

    * cT3-cT4
    * Grade Group 4 or 5
    * PSA > 40 ng/mL\
* Willing and able to undergo prostate MRI at baseline, with a measurable prostate lesion present.
* Planning to undergo radical prostatectomy as primary treatment for localized prostate cancer.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Adequate bone marrow and organ function as defined below:

  * Leukocytes ≥ 3.0 K/cumm
  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Estimated glomerular filtration rate eGFR ≥ 30 mL/min/1.73m^2
* Agreement to adhere to Lifestyle Considerations throughout study duration
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Current or previous treatment with SGLT2i or thiazolidinedione.
* Currently receiving regularly scheduled systemic steroids in the form of prednisone or dexamethasone (more than 10 mg prednisone daily or equivalent). Topical steroid ointments or creams for occasional skin rash is allowed.
* A history of other malignancy with the exceptions of malignancies for which all treatment was completed at least 2 years before registration with no evidence of disease and locally treated skin squamous or basal cell carcinoma.
* History of stroke or transient ischemic attack in the last 5 years.
* Patients with type 1 diabetes mellitus will be excluded or patients with insulin-requiring diabetes mellitus will be excluded. Only patients with well-controlled type 2 diabetes mellitus will be allowed.
* Screening HbA1c > 10%, unless approved by endocrinologist.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to dapagliflozin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, peripheral arterial disease, ketoacidosis, severe kidney disease (estimated glomerular filtration rate eGFR < 30 mL/min/1.73m2), symptomatic hypotension, and chronic/frequent urinary tract infections or yeast infections.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.
* Any evidence of pelvic instrumentation (i.e. hip arthroplasty) that would obscure and/or limit prostate MRI evaluation at the discretion of the investigator, or any type of medical device that would be incompatible with MRI imaging.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of toxicities related to dapagliflozin as measured by CTCAE v 5.0 | From cycle 1 day 1 (the cycle is 28 days in length) through 30 days after prostatectomy (approximately day 64)
Proportion of patients who are able to successfully complete at least 80% of the planned dapagliflozin doses and undergo radical prostatectomy | At approximately 6 weeks
  The study will be feasible if at least 19 of the 24 enrolled subjects are able to complete at least 80% of the planned dapagliflozin doses and undergo radical prostatectomy as scheduled.

SECONDARY OUTCOMES:
MRI quantified change in tumor size from screening to post-treatment | At the time of pre-operative prostate MRI (estimated to be at week 6)
Degree of tumor necrosis/shrinking | From screening to time of radical prostatectomy (estimated to be at week 6)
Change in plasma glucose | From screening to day 29
Change in C-peptide | From screening to day 29
Change in HbA1C | From screening to day 29
Change in glucagon | From screening to day 29

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Reimers, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu